CLINICAL TRIAL: NCT02611544
Title: Investigation of Three Approaches to Address Fear of Recurrence Among Breast Cancer Survivors: A Randomized Clinical Pilot Trial
Brief Title: Investigation of Three Approaches to Address Fear of Recurrence Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Shelley Johns, Assistant Professor of Medicine, Research Scientist, Indiana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IUSCC-0563
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Breast Neoplasms; Breast Cancer; Breast Carcinoma; Malignant Neoplasm of Breast; Cancer of Breast; Mammary Neoplasm, Human; Human Mammary Carcinoma; Malignant Tumor of Breast; Mammary Cancer; Mammary Carcinoma; Anxiety; Fear; Neoplasm Remission, Spontaneous; Spontaneous Neoplasm Regression; Regression, Spontaneous Neoplasm; Remission, Spontaneous Neoplasm; Spontaneous Neoplasm Remission
Keywords: Fear of Cancer Recurrence; Fear of Cancer Return; Breast Cancer Survivor; Breast Cancer Remission
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Neoplasm Regression, Spontaneous | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Masking Description: Participants were blinded to study hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance and Commitment Therapy (Active Comparator): 6 weeks, the ACT group will meet weekly for 2 hours at one of three facilities.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Survivorship Education (Active Comparator): 6 weeks, SE group will meet weekly for 2 hours at one of three facilities.
  Interventions: Behavioral: Survivorship Education
- Enhanced Usual Care (Active Comparator): Continue to meet with their health care team + receive a variety of readings at each data collection point on coping with common survivorship concerns, including a booklet from the National Cancer Institute entitled "Facing Forward: Life After Cancer Treatment."
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — 6-week ACT intervention group (n=33)
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy
Behavioral: Survivorship Education — 6-week survivorship education group (SE; n=32)
  Other Names: SE
  Arms: Survivorship Education
Behavioral: Enhanced Usual Care — enhanced usual care (EUC; n=26)
  Other Names: EUC
  Arms: Enhanced Usual Care

SUMMARY:
Fear of cancer recurrence (FCR) is one of the most prevalent, persistent, and disruptive sources of distress for adult cancer survivors. Prevalence rates for FCR have been estimated at up to 89%, with approximately half of cancer survivors reporting clinically significant levels of FCR. Despite the recognized prevalence, persistence, and suffering associated with FCR, effective and accessible treatments for FCR are lacking and urgently needed. Our long-term goal is to develop, evaluate, and implement effective behavioral interventions for cancer survivors suffering with FCR.

DETAILED DESCRIPTION:
The proposed randomized pilot study will assess the effects of a novel therapeutic intervention-Acceptance and Commitment Therapy (ACT)-for breast cancer survivors (BCS) with clinically-significant FCR. ACT is a spiritually-sensitive behavioral therapy that has shown efficacy in the treatment of anxiety in non-cancer populations, and preliminary efficacy in improving a variety of outcomes among adults with cancer. ACT uses mindfulness and acceptance processes, along with committed behavior change in service of an individual's deeply held values to enhance psychological flexibility and encourage adaptive coping with life challenges, such as cancer.

The primary objective of the proposed 3-arm randomized controlled pilot trial is to assess the feasibility/acceptability and determine preliminary effect size estimates of ACT in preparation for a fully-powered efficacy trial. To allow for potential drop out (15% attrition) and ensure we have a minimum of 78 completers through the end of the trial, we will enroll approximately 91 BCS with clinically significant FCR (defined by score ≥ 13 on Fears of Cancer Recurrence Inventory-Short Form). Participants will be randomized to one of three groups: (1) a 6-week ACT intervention group (n=26); (2) a 6-week survivorship education group (SE; n=26); or (3) enhanced usual care (EUC; n=26). The impact of ACT, SE, and EUC on survivors' FCR and associated psychological, spiritual, and biological (telomere length) outcomes will be examined at baseline (T1), post-intervention (T2), and at 1-month (T3) and 6-month follow-up (T4) with the following specific aims:

Aim 1: Evaluate feasibility and acceptability of ACT, SE, and EUC according to the:

1. Percentage of eligible BCS who consent to participate in the trial;
2. Attendance rate across 6 sessions of ACT and SE;
3. Retention rate through T4 in the ACT, SE, and EUC arms;
4. Mean ratings across groups for intervention satisfaction and helpfulness for managing FCR.

Aim 2: Determine pairwise effect size estimates of ACT, SE, and EUC effects at each time point (T2, T3, T4) adjusted for T1 on the:

1. Primary outcome: reducing FCR;
2. Secondary psychological outcomes: cancer-related experiential avoidance, cognitive avoidance, anxiety, depression, post-traumatic stress symptoms, vitality, breast cancer self-efficacy, and quality of life;
3. Secondary spiritual outcomes: spiritual well-being and mindfulness;
4. Secondary biological outcome: telomere length.

ELIGIBILITY:
Inclusion Criteria: Participants in this study will be eligible if they are:

1. ≥18 years old,
2. have been diagnosed with non-metastatic breast cancer (stages I-III),
3. have completed curative treatment for breast cancer,
4. have not experienced a cancer recurrence, and
5. report a clinically significant level of FCR (Fear of Cancer Recurrence Inventory-Short Form score of ≥ 13)

Exclusion Criteria: Participants in this study will be ineligible if they are:

1. severe depression (PHQ-8 score of ≥ 20),
2. past participation in ACT or formal mindfulness training, and
3. limited English proficiency.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fear of recurrence (FCR) at Post-Intervention, 1-month, and 6-month follow-up as assessed by Fear of Cancer Recurrence Inventory (FCRI). | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Fear of Cancer Recurrence Inventory (FCRI)

SECONDARY OUTCOMES:
Change from baseline in fear of recurrence (FCR) at Post-Intervention, 1-month, and 6-month follow-up as assessed by Concerns about Recurrence Scale (CARS). | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Concerns about Recurrence Scale (CARS)
Change from baseline in cancer-related avoidant coping at Post-Intervention, 1-month, and 6-month follow-up as assessed by Acceptance & Action Questionnaire-Cancer | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Acceptance & Action Questionnaire-Cancer
Change from baseline in anxiety at Post-Intervention, 1-month, and 6-month follow-up as assessed Generalized Anxiety Disorder Scale (GAD-7). | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Generalized Anxiety Disorder Scale (GAD-7)
Change from baseline in depression at Post-Intervention, 1-month, and 6-month follow-up as assessed by as measured by Patient Health Questionnaire Depression Scale (PHQ-8). | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Patient Health Questionnaire Depression Scale (PHQ-8)
Change from baseline in post-traumatic stress symptoms at Post-Intervention, 1-month, and 6-month follow-up as assessed by Impact of Events Scale-Revised (IES-R). | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Impact of Events Scale-Revised (IES-R)
Change from baseline in vitality at Post-Intervention, 1-month, and 6-month follow-up as assessed by Short Form(SF)-36 Vitality Scale. | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Short Form(SF)-36 Vitality Scale
Change from baseline in Breast Cancer Self-Efficacy at Post-Intervention, 1-month, and 6-month follow-up as assessed by Breast Cancer Self-Efficacy Scale | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Breast Cancer Self-Efficacy Scale
Change from baseline in quality of life at Post-Intervention, 1-month, and 6-month follow-up as assessed by 10-item PROMIS Global Health Scale | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by PROMIS Global Health Scale
Change from baseline in spiritual well-being at Post-Intervention, 1-month, and 6-month follow-up as assessed by Functional Assessment of Chronic Illness Therapy-Spiritual Well-being (FACIT-Sp) scale | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Functional Assessment of Chronic Illness Therapy- Spiritual Well-being (FACIT-Sp) scale
Change from baseline in mindfulness at Post-Intervention, 1-month, and 6-month follow-up as assessed by Five Facet Mindfulness Questionnaire-Short Form | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by Five Facet Mindfulness Questionnaire-Short Form
Change from baseline in telomere length at Post-Intervention, 1-month, and 6-month follow-up as assessed by quantitative telomere length. | Baseline (T1), post-intervention/6-weeks (T2), 1-month (T3), and 6-month follow-up (T4)
  As measured by quantitative telomere length.
Intervention ratings for satisfaction and helpfulness at Post-Intervention as assessed by a 5-item investigator-created measure. | post-intervention/6-weeks (T2)
  As measured by a 5-item investigator-created measure of intervention satisfaction and helpfulness

CONTACTS AND LOCATIONS:
Overall Officials: Shelley A Johns, PsyD, Principal Investigator — Indiana University School of Medicine; Regenstrief Institute, Inc.
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Koch L, Jansen L, Brenner H, Arndt V. Fear of recurrence and disease progression in long-term (>/= 5 years) cancer survivors--a systematic review of quantitative studies. Psychooncology. 2013 Jan;22(1):1-11. doi: 10.1002/pon.3022. Epub 2012 Jan 10. PMID 22232030
- [Background] Vickberg SM. The Concerns About Recurrence Scale (CARS): a systematic measure of women's fears about the possibility of breast cancer recurrence. Ann Behav Med. 2003 Winter;25(1):16-24. doi: 10.1207/S15324796ABM2501_03. PMID 12581932
- [Background] Needham BL, Mezuk B, Bareis N, Lin J, Blackburn EH, Epel ES. Depression, anxiety and telomere length in young adults: evidence from the National Health and Nutrition Examination Survey. Mol Psychiatry. 2015 Apr;20(4):520-8. doi: 10.1038/mp.2014.89. Epub 2014 Sep 2. PMID 25178165
- [Background] Duggan C, Risques R, Alfano C, Prunkard D, Imayama I, Holte S, Baumgartner K, Baumgartner R, Bernstein L, Ballard-Barbash R, Rabinovitch P, McTiernan A. Change in peripheral blood leukocyte telomere length and mortality in breast cancer survivors. J Natl Cancer Inst. 2014 Apr;106(4):dju035. doi: 10.1093/jnci/dju035. Epub 2014 Mar 13. PMID 24627273
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Lebel S, Maheu C, Lefebvre M, Secord S, Courbasson C, Singh M, Jolicoeur L, Benea A, Harris C, Fung MF, Rosberger Z, Catton P. Addressing fear of cancer recurrence among women with cancer: a feasibility and preliminary outcome study. J Cancer Surviv. 2014 Sep;8(3):485-96. doi: 10.1007/s11764-014-0357-3. Epub 2014 Apr 23. PMID 24756313
- [Background] Butow PN, Bell ML, Smith AB, Fardell JE, Thewes B, Turner J, Gilchrist J, Beith J, Girgis A, Sharpe L, Shih S, Mihalopoulos C; members of the Conquer Fear Authorship Group. Conquer fear: protocol of a randomised controlled trial of a psychological intervention to reduce fear of cancer recurrence. BMC Cancer. 2013 Apr 23;13:201. doi: 10.1186/1471-2407-13-201. PMID 23617696
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Feros DL, Lane L, Ciarrochi J, Blackledge JT. Acceptance and Commitment Therapy (ACT) for improving the lives of cancer patients: a preliminary study. Psychooncology. 2013 Feb;22(2):459-64. doi: 10.1002/pon.2083. Epub 2011 Oct 6. PMID 23382134
- [Background] Hulbert-Williams NJ, Storey L, Wilson KG. Psychological interventions for patients with cancer: psychological flexibility and the potential utility of Acceptance and Commitment Therapy. Eur J Cancer Care (Engl). 2015;24(1):15-27. doi: 10.1111/ecc.12223. Epub 2014 Aug 6. PMID 25100576
- [Background] Johns SA, Brown LF, Beck-Coon K, Monahan PO, Tong Y, Kroenke K. Randomized controlled pilot study of mindfulness-based stress reduction for persistently fatigued cancer survivors. Psychooncology. 2015 Aug;24(8):885-93. doi: 10.1002/pon.3648. Epub 2014 Aug 17. PMID 25132206
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Fischer D, Stewart AL, Bloch DA, Lorig K, Laurent D, Holman H. Capturing the patient's view of change as a clinical outcome measure. JAMA. 1999 Sep 22-29;282(12):1157-62. doi: 10.1001/jama.282.12.1157. PMID 10501119
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Watson M, Law, M.G., Santos, M.D., Greer, S., Baruch, J., Bliss, J. . The Mini-MAC. J Psychosoc Oncol. 1994;12(3):33-46.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Weiss D, Marmar C. The Impact of Event Scale-Revised. In: Wilson J, Keane T, editors. Assessing psychological trauma and PTSD: A practicioner's handbook. New York: Guilford Press; 1997. p. 399-411.
- [Background] Ware J, Snow K, Kosinski M. SF-36 healthy survey manual and interpretation guide. Lincoln, RI: Quality Metric Inc.; 1993.
- [Background] Champion VL, Ziner KW, Monahan PO, Stump TE, Cella D, Smith LG, Bell CJ, Von Ah D, Sledge GW. Development and psychometric testing of a breast cancer survivor self-efficacy scale. Oncol Nurs Forum. 2013 Nov;40(6):E403-10. doi: 10.1188/13.ONF.E403-E410. PMID 24161644
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809